CLINICAL TRIAL: NCT00779896
Title: Tazarotene 0.1% Cream For the Treatment of Cutaneous T-Cell Lymphoma: A Prospective Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Responsible Party: Dr. David Roberger, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: McG 0722
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Cutaneous T-Cell Lymphoma
Keywords: To evaluate therapeutic potential of tazarotene 0.1% cream for the treatment of Stage I-IIA CTCL. Patients with Stage I-IIA disease are enrolled into the study; Stage I-IIA disease CTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — tazarotene; tazarotenic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tazarotene — Topical 0.1 cream - apply to lesions on alternate days and at 2 week interval increase to once-daily application, if tolerated.
  Other Names: Tazorac (trademark name); Tazarotenic Acid

SUMMARY:
This is an open label, prospective study to evaluate therapeutic potential of Tazarotene 0.1% cream for the treatment of Stage I-IIA CTCL. Patients with Stage I-IIA disease are enrolled into the study. Tazarotene will be used for up to 24 weeks and patients will be followed for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage I-IIA CTCL must be at least 18 years of age with a skin biopsy prior to enrolment confirming the diagnosis of mycosis fungoides.

Exclusion Criteria:

* Patients with Stage >IIA CTCL at the time of enrolment
* Women who are pregnant or planning to get pregnant, or unable/unwilling to use adequate contraception
* Patients who were treated with topical retinoid therapy in the past 3 months
* Patients who received any systemic CTCL therapy or systemic corticosteroid therapy within 30 days of the study start date
* Patients who were treated with systemic isotretinoin or bexarotene within 3 months prior to the study start date, systemic acitretin within 2 years prior to study start date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Partial response (PR) is defined as some improvement (25%-50%);significant evidence of disease remains or disease has not changed from baseline condition (<25%);no new clinically abnormal(>1.5 cm)lymph nodes,<25% progression of existence

CONTACTS AND LOCATIONS:
Overall Officials: David Roberge, Principal Investigator — Montreal General Hospital
Locations (1):
- McGill University, Montreal, Quebec, Canada